CLINICAL TRIAL: NCT03979378
Title: Treatment of Ectopic Calcification / Ossification With Sodium Thiosulfate (CATSSO)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: CATSSO
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Sodium Thiosulfate; Ectopic Ossification
MeSH Terms: conditions — Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Ectopic calcification and ossification complicate many diseases, which are rare for the most part. These calcifications (or ossifications) are generally classified according to their apparent formation mechanism. Even if very different diseases can be at the origin, these calcifications (or ossifications) have as common points: an unknown physiopathology, a composition of calcium pyrophosphate for the most part and l no curative treatment validated to date.

Indeed, although several reported cases suggest the potential efficacy of different treatments , none of these treatments is currently recognized as effective because of the absence of confirmation data or because of contradictory results.

Sodium thiosulfate (STS) has been used for a long time as an antidote to cyanide poisoning and as a protective agent against cytotoxic side effects such as ifosphamide. More recently, STS has been reported in the treatment of renal calcification. vascular or even subcutaneous. First prospective studies on animal models and in humans seem to confirm the interest of this product in the treatment of these abnormal calcifications.

For several months, a magistral preparation in the form of ointment based on STS has been developed by the pharmacy of Limoges University Hospital in order to combine the local effect of STS while avoiding the side effects of an administration of this treatment by systemic way. The first uses of this preparation appear promising and some preliminary results have already been published. The benefit / risk ratio of this approach seems to be advantageous for clinicians since preparations whose composition is close are currently validated by the FDA and the World Health Organisation for the treatment of benign pathologies such as cutaneous dermatophytes or pityriasis versicolor.

ELIGIBILITY:
Inclusion Criteria:

* any patient treated with sodium thiosulfate dermally provided by the pharmacy of Limoges University Hospital.
* availability of an objective imaging evaluation to compare the volume or surface of calcifications (or ossifications) treated (on two orthogonal incidences) before and after 6 months of treatment application.
* consent to participation in the study signed by the patient or by one of the holders of parental authority in the case of a minor patient.

Exclusion Criteria:

* calcification with concomitant cutaneous rupture which can allow an externalization of the calcium material by mechanical effects.
* Patient with calcification secondary to one of the following pathologies:
* diabetes
* chronic renal failure
* iatrogenic origin

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with ectopic calcification / ossification
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Calcification/Ossification volume | Month 6
  Percentage decrease in the volume or surface area of calcifications (or ossification) treated on imaging of the same type performed before and 6 months after dermal STS use.

SECONDARY OUTCOMES:
Change in aesthetic evolution from baseline at 6 month | Day 0, Month 6
  aesthetic evolution on picture
Change in pain from baseline at 6 month | Day 0, Month 6
  Evaluation of pain with scale VAE (visual analog evaluation)
Change of the quality of life from baseline at 6 month | Day 0, Month 6
  evolution of the quality of life with Skindex scale
local or general side effects | Month 6
  Number and nature of local or general side effects

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Grenoble university hospital, Grenoble
  - Kremlin Bicetre Hospital, Le Kremlin-Bicêtre
  - CHU de Limoges, Limoges
  - HEGP, Paris
  - Lariboisière Hospital, Paris
  - Necker Hospital, Paris
  - Robert Debré Hospital, Paris